CLINICAL TRIAL: NCT01646437
Title: The International Polycap Study 3 (TIPS-3) is a Randomized Double-blind Placebo-controlled Trial for the Evaluation of a Polycap, Low Dose Aspirin and Vitamin D Supplementation in Primary Prevention
Brief Title: The International Polycap Study 3 (TIPS-3)
Acronym: TIPS-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Cadila Pharnmaceuticals (Industry); Wellcome Trust (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Principal Investigator, Salim Yusuf's office, Executive Director - Population Health Research Institute, Professor of Medicine - McMaster University, Population Health Research Institute
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TIPS-3
Record Dates: First submitted 2012-07-10; First posted 2012-07-20 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Cardiovascular Disease; Fractures; Cancers
MeSH Terms: conditions — Cardiovascular Diseases; Fractures, Bone; Neoplasms | interventions — Aspirin; Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Polycap vs. matching placebo (Experimental): Polycap is a once daily capsule containing thiazide (25mg), atenolol (100mg), ramipril (10mg) and simvastatin (40mg) vs. matching placebo
  Interventions: Drug: Polycap; Drug: Matching Placebo
- Aspirin vs. matching placebo (Experimental): Once daily 75mg tablet of Aspirin vs. matching placebo
  Interventions: Drug: Aspirin; Drug: Matching Placebo
- Vitamin D vs. matching placebo (Experimental): Monthly oral dosage of 60,000IU vs. matching placebo
  Interventions: Drug: Vitamin D; Drug: Matching Placebo

INTERVENTIONS:
Drug: Polycap — Polycap (thiazide 25mg, atenolol 100mg, ramipril 10mg, simvastatin 40mg) taken once daily
  Arms: Polycap vs. matching placebo
Drug: Aspirin — 75 mg daily
  Other Names: enteric coated aspirin
  Arms: Aspirin vs. matching placebo
Drug: Vitamin D — 60,000 IU monthly
  Other Names: cholecalciferol
  Arms: Vitamin D vs. matching placebo
Drug: Matching Placebo — Matching Placebo

SUMMARY:
The randomized 2x2x2 factorial design placebo controlled trial will enroll 5000 participants (women 60 years or older and men 55 years or older) without known heart disease or prior stroke and without a clear indication or contraindication to any of the study medications. Eligible and consenting individuals will be randomized to receive either the active study medications or placebo (dummy pills) and will be monitored for an average of 5 years. The study will include people from at 10 countries, will be conducted by an international group of scientists and physicians and will be coordinated by the Population Health Research Institute at Hamilton Health Sciences.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD), cancers and osteoporosis collectively make up the largest disease burden globally. CVD is the major cause of death and disability and affects about half of the population over their lifetimes. Cancers are a leading cause of death and it accounts for 13.0% of all deaths. The commonest forms include lung, breast, prostate, colorectum, stomach and liver cancer. It is estimated that over 200 hundred million people worldwide are living with osteoporosis. This is the underlying pathologic predisposition to fractures of the hip, vertebral body, and distal forearm. CVD, cancers and osteoporotic fractures increase with age and so their burden is expected to substantially increase over the next few decades. Simple, safe and effective preventive strategies which can reduce the incidence and prevalence of these 3 diseases are therefore urgently needed

It is suggested that this polypill could be given to all individuals with a CVD event as well as to anyone over 55 years (primary prevention) without the need for any measurement of risk factors. The polypill contains 3 blood pressure lowing medications and a statin in a single tablet. This includes hydrochlorothiazide (25 mg), atenolol (100 mg), ramipril (10 mg) and simvastatin (40 mg). In addition, to the polypill (Polycap), participants will be randomized to receive aspirin (75mg) and vitamin D (60,000 IU monthly). This factorial design on 3 distinct treatment arms which could reduce CVD, fractures and cancers could have large implications for the prevention of several of the important chronic diseases in middle and old age, using safe and inexpensive medications/supplements.

ELIGIBILITY:
Inclusion Criteria:

* Men aged ≥ 50 years and women aged ≥ 55 years with an INTERHEART risk score ≥ 10 OR men and women aged ≥ 65 years with an INTERHEART risk score of ≥5.
* Provision of informed consent

Exclusion Criteria

* Participants with a clear clinical indication, contraindication, preference for or intolerance to statin, beta blocker (e.g. bradycardia), ACE inhibitor, diuretic, aspirin or clopidogrel in the judgment of the physician.
* Regular use of vitamin D at doses higher than 400 IU per day.
* Hypercalcemia, hyperparathyroidism, osteomalacia or other contraindication or indication for vitamin D therapy.
* Peptic ulcer disease, frequent dyspepsia or bleeding.
* Expected long term use of anticoagulants
* Known vascular disease. (e.g., Stroke, TIA, Angina, MI, ACS, PVD including claudication and amputation).
* Mean systolic BP (using 2 automatic readings) below 120 mm Hg at run-in.
* Symptomatic hypotension (e.g., dizziness with SBP <110 mm Hg systolic) during the run-in phase.
* Chronic liver disease or abnormal liver function, i.e. ALT or AST > 3 x ULN.
* Inflammatory muscle disease (such as dermatomyositis or polymyositis) or creatine kinase (CK) > 3 x ULN.
* Severe renal impairment (serum creatinine >264 µmol/L).
* History of malignancy affecting any organ system, except basal cell carcinoma of the skin, within the previous 5 years.
* Other serious condition(s) likely to interfere with study participation or with the ability to complete the trial.
* Concurrent use of any experimental pharmacological agent.
* Inability to attend follow-up as required by the protocol for at least 5 years.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7793 (Actual)
Dates: Start 2012-06; Primary Completion 2020-06-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Polycap Primary Objective | Participants will be followed for an average of 4.25 years
  To determine whether the Polycap reduces the risk of the composite outcome of CVD events which includes major CVD (CV death, non-fatal stroke, non-fatal MI), plus heart failure, resuscitated cardiac arrest, or arterial revascularization compared to placebo.
Aspirin Primary Objective | Participants will be followed for an average of 4.25 years
  To determine whether aspirin reduces the risk of composite outcome of major CV events (CV death, non-fatal MI or non-fatal stroke,) compared to its placebo.
Vitamin D Primary Objective | Participants will be followed for an average of 4.25 years
  To determine whether vitamin D reduces the risk of fractures compared to its placebo.
Combined Effects of Polycap and Aspirin on CVD Events | Participants will be followed for an average of 4.25 years
  To determine the combined effect of aspirin and the Polycap (i.e. double treatment) on major CV events (CV death, non-fatal MI or non-fatal stroke), heart failure, resuscitated cardiac arrest, or arterial revascularization compared to double-placebo.

SECONDARY OUTCOMES:
Polycap Secondary Objective | Participants will be followed for an average of 4.25 years
  To determine whether the Polycap reduces the risk of the composite of CV death, non-fatal stroke, and non-fatal MI compared to its placebo.To determine whether the Polycap reduces the risk of the composite outcome of major CVD (CV death, non- fatal stroke, non-fatal myocardial infarction [MI]), heart failure, resuscitated cardiac arrest, arterial revascularization, or angina with evidence of ischemia.
Aspirin Secondary Objective | Participants will be followed for an average of 4.25 years
  To determine whether a daily aspirin reduces the risk of the composite outcome of major CV events (CV death, non-fatal MI or non-fatal stroke) and cancers compared to its placebo.
Vitamin D Secondary Objective | Participants will be followed for an average of 4.25 years
  To determine whether vitamin D reduces the risk of the composite outcome of CV events, fractures and cancers, and the risk of falls compared to its placebo.
Combined Effects of Polycap and Aspirin on CVD Events Secondary Outcome A | Participants will be followed for an average of 4.25 years
  To determine whether the Polycap and aspirin reduces the risk of the composite of CV death, non-fatal stroke, and non-fatal MI compared to double placebo.
Combined Effects of Polycap and Aspirin on CVD Events Secondary Outcome B | Participants will be followed for an average of 4.25 years
  To determine whether the Polycap and aspirin reduces the risk of the composite outcome of major CVD (CV death, non- fatal stroke, non-fatal myocardial infarction [MI]), heart failure, resuscitated cardiac arrest, arterial revascularization, or angina with evidence of ischemia, compared to double-placebo

OTHER OUTCOMES:
Total mortality | Participants will be followed for an average of 4.25 years
  To assess the effect of each of the 3 treatments on total mortality.
Incident and recurrent CV events | Participants will be followed for an average of 4.25 years
  To determine whether the Polycap reduces the risk of incident and recurrent CV events (which is comprised of major CVD (CV death, non- fatal stroke, non-fatal myocardial infarction [MI]), plus heart failure, resuscitated cardiac arrest or arterial revascularization)).
Long term safety | Participants will be followed for an average of 4.25 years
  To assess the long-term safety of each treatment (Polycap, Aspirin or Vitamin D) versus their respective placebo on safety and tolerability.
Visual acuity | Participants will be followed for an average of 4.25 years
  To assess the effect of the Polycap and Aspirin on visual acuity change from baseline and onset of age-related macular degeneration.
Cognitive Function | Participants will be followed for an average of 4.25 years
  To assess the effect of each of the 3 treatments on cognitive function
Health Economics | Participants will be followed for an average of 4.25 years
  To assess the economic impact of the Polycap

CONTACTS AND LOCATIONS:
Overall Officials: Salim Yusuf, Principal Investigator — Population Health Research Institute; Prem Pais, Principal Investigator — St. John's Research Institute
Locations (9):
- Eminence, Dhaka, Bangladesh
- Hamilton Health Sciences, Hamilton, Ontario, Canada
- Fundaction Oftamologica De Santander (FOSCAL), Bucaramanga, Colombia
- St. John's Medical College Hospital, Bangalore, India
- Harapan Kita Hopsital, Jakarta, Indonesia
- Universiti Teknologi MARA (UiTM), Shah Alam, Selangor, Malaysia
- Adult Medicine & Medical Research Unit, Philippine General Hospital, Manila, Philippines
- Pamoja Tunaweza Women's Centre, Moshi, Tanzania
- Fattouma Bourguiba University Hospital, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Joseph P, Pais P, Gao P, Teo K, Xavier D, Lopez-Jaramillo P, Yusoff K, Santoso A, Gamra H, Talukder SH, Christou C, Dagenais G, Tyrwhitt J, Bosch J, Dans A, Yusuf S; International Polycap Study (TIPS)-3 Investigators. Vitamin D supplementation and adverse skeletal and non-skeletal outcomes in individuals at increased cardiovascular risk: Results from the International Polycap Study (TIPS)-3 randomized controlled trial. Nutr Metab Cardiovasc Dis. 2023 Feb;33(2):434-440. doi: 10.1016/j.numecd.2022.11.001. Epub 2022 Nov 15. PMID 36604262
- [Derived] Yusuf S, Joseph P, Dans A, Gao P, Teo K, Xavier D, Lopez-Jaramillo P, Yusoff K, Santoso A, Gamra H, Talukder S, Christou C, Girish P, Yeates K, Xavier F, Dagenais G, Rocha C, McCready T, Tyrwhitt J, Bosch J, Pais P; International Polycap Study 3 Investigators. Polypill with or without Aspirin in Persons without Cardiovascular Disease. N Engl J Med. 2021 Jan 21;384(3):216-228. doi: 10.1056/NEJMoa2028220. Epub 2020 Nov 13. PMID 33186492
- [Derived] Joseph P, Pais P, Dans AL, Bosch J, Xavier D, Lopez-Jaramillo P, Yusoff K, Santoso A, Talukder S, Gamra H, Yeates K, Lopez PC, Tyrwhitt J, Gao P, Teo K, Yusuf S; TIPS-3 Investigators. The International Polycap Study-3 (TIPS-3): Design, baseline characteristics and challenges in conduct. Am Heart J. 2018 Dec;206:72-79. doi: 10.1016/j.ahj.2018.07.012. Epub 2018 Aug 2. PMID 30342297